CLINICAL TRIAL: NCT00241085
Title: A Multi-center, Double Blind, Randomized, Parallel Group Study to Evaluate the Effects of Valsartan on Proteinuria in Hypertensive Subjects With Type 2 Diabetes Mellitus
Brief Title: Effect of Valsartan on Proteinuria in Patients With Hypertension and Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489A2417
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-06

CONDITIONS: PROTEINURIA; Hypertension; Type 2 Diabetes
Keywords: proteinuria; hypertension; valsartan; type 2 diabetes
MeSH Terms: conditions — Proteinuria; Hypertension; Diabetes Mellitus, Type 2 | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
This is a study of whether valsartan affects levels of proteinuria in patients with type 2 diabetes and hypertension.

ELIGIBILITY:
Inclusion Criteria:

- Mild to moderate hypertension, Mild renal dysfunction, Type 2 diabetes,

Exclusion Criteria:

Pregnant or breast feeding, Type 1 diabetes

Other protocol criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2002-11; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urinary protein excretion after 30 weeks

SECONDARY OUTCOMES:
Change from baseline in circulating markers of blood vessel inflammation, insulin resistance, serum creatinine, diabetic control, and proportion of patients who return to normalization of protein excretion after 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Weir MR, Hollenberg NK, Zappe DH, Meng X, Parving HH, Viberti G, Remuzzi G. Antihypertensive effects of double the maximum dose of valsartan in African-American patients with type 2 diabetes mellitus and albuminuria. J Hypertens. 2010 Jan;28(1):186-93. doi: 10.1097/HJH.0b013e328332bd61. PMID 19809363